CLINICAL TRIAL: NCT02916030
Title: Vitamin D and Stroke: A Comparative Study to Risk Factors and Stroke Type
Brief Title: Vitamin D and Stroke
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Professor (Anesthesiology and Critical Care)- College of Medicine-Assiut University, Assiut University
Other Study IDs: IRB0000871535
Record Dates: First submitted 2016-09-17; First posted 2016-09-27 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Stroke
Keywords: Vitamin D; Stroke; Parathormone
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1 (hemorrhagic stroke): All participants will be subjected to thorough history taking, full clinical and neurological examination. Stroke subtype will be classified according to the criteria of Trial of Org 10172 in acute Stroke Treatment (TOAST) classification.
  Interventions: Dietary Supplement: Vit D
- Group 2 (Ischemic stroke): All participants will be subjected to thorough history taking, full clinical and neurological examination. Stroke subtype will be classified according to the criteria of Trial of Org 10172 in acute Stroke Treatment (TOAST) classification.
  Interventions: Dietary Supplement: Vit D

INTERVENTIONS:
Dietary Supplement: Vit D — It is to examine the relationship between serum 25 (OH) D levels and Stroke either ischemic or hemorrhagic types

SUMMARY:
Stroke remains one of the most devastating neurological diseases, often causing death, or gross physical impairment. It is the second most common cause of death worldwide and a major cause of acquired disability in adults.Vitamin D deficiency has been reported to contribute to the risk of cardiovascular disease especially stroke.

DETAILED DESCRIPTION:
This case -control observational prospective study will conducted on fifty patients with first -ever acute onset stroke within seven days (25 patients with hemorrhagic stroke and 25 patients with ischemic stroke )

ELIGIBILITY:
Inclusion Criteria:

* Onset is within one week
* Confirmed stroke by brain CAT and / or MRI scan either haemorrhage or infarction

Exclusion Criteria:

* Cognitive and mental changes
* Recurrent stroke
* Hepatic and renal impairment
* Endocrinal diseases
* Steroid therapy
* Vitamin D or Ca supplementation
* Previous fractures
* Bone diseases
* brain neoplasm,
* Autoimmune diseases
* History of acute and chronic inflammatory diseases
* Malignancy,
* Trauma
* Surgery
* Acute vascular diseases that occurred within four weeks prior the onset of stroke
* History myocardial infarction ˂3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with first -ever acute onset stroke within seven days
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2017-01-03 (Actual)

PRIMARY OUTCOMES:
serum 25 (OH) D levels | Within the first 24 hours
  serum 25 (OH) D levels

SECONDARY OUTCOMES:
Stroke severity | Within the first 24 hours
  Stroke severity will be assessed by Scandinavian Stroke scale Stroke (SSS)
Stroke etiology | Within the first 24 hours
Stroke risk factors | Within the first 24 hours
Stroke subtypes | Within the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: sayed abd elshafy, MD, Principal Investigator — associate professor of anesthesia and critical care
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided